CLINICAL TRIAL: NCT03739411
Title: Pilot Study of Safety and Feasibility of Acquiring Hyperpolarized Imaging in Patients With Gliomas
Brief Title: Hyperpolarized Imaging in Diagnosing Participants With Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Susan Chang (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Susan Chang, Professor in Residence and Vice Chair of Neurological Surgery, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13106; NCI-2018-00939 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); R01CA109767 (NIH); R01CA273028 (NIH); 2P50CA097257 (NIH)
Record Dates: First submitted 2018-05-29; First posted 2018-11-13 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort I (Hyperpolarized C13, MRI) (Experimental): Participants receive hyperpolarized carbon C 13 pyruvate intravenously IV and undergo MRI. The second hyperpolarized 13 C injection/imaging will be started approximately 15 to 60 minutes after the first injection for those who are willing to receive two 13 C injections
  Interventions: Radiation: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Imaging
- Cohort II (Hyperpolarized C13, MRI) (Experimental): Participants receive hyperpolarized carbon C 13 pyruvate IV and undergo MRI before treatment and 4 weeks after completion of cancer therapy given outside of this study.
  Interventions: Radiation: Hyperpolarized Carbon C 13 Pyruvate; Procedure: Magnetic Resonance Imaging; Radiation: Radiation Therapy; Drug: Chemotherapy

INTERVENTIONS:
Radiation: Hyperpolarized Carbon C 13 Pyruvate — Given IV
  Other Names: Hyperpolarized Pyruvate (13C)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MRI; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Radiation: Radiation Therapy — Undergo radiation therapy for cancer outside of this study.
  Other Names: Radiotherapeutics; Radiotherapy
  Arms: Cohort II (Hyperpolarized C13, MRI)
Drug: Chemotherapy — Undergo chemotherapy for cancer outside of this study.
  Arms: Cohort II (Hyperpolarized C13, MRI)

SUMMARY:
This pilot trial studies the side effects of hyperpolarized carbon C 13 pyruvate magnetic resonance imaging (MRI) in diagnosing participants with glioma. Diagnostic procedures, such as hyperpolarized carbon C 13 pyruvate MRI, may help find and diagnose glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and feasibility of hyperpolarized 13C MR metabolic imaging as a new and unique tool for evaluating tumor burden and detecting early response to therapy in participants with glioma.

II. To define the most appropriate imaging parameters for obtaining hyperpolarized 13C data from the brain, one hundred participants with evidence of residual disease from a prior MRI examination will have hyperpolarized metabolic imaging after receiving one or two injections of hyperpolarized 13 C pyruvate. For participants who are willing to receive two injections, the 2nd injection will be used to assess reproducibility, evaluate the performance of new acquisition methods, or compare metabolism between [1-13C]pyruvate and [213C]pyruvate.

III. To establish the time course of changes in hyperpolarized pyruvate and lactate peaks on a voxel by voxel basis from the dynamic hyperpolarized data after the injection(s) of hyperpolarized 13C pyruvate. Twenty participants will be studied before and after treatment with treatment in order to determine the time course of delivery of 13C pyruvate and the location of maximum pyruvate and lactate or glutamate signals in normal brain and in the region of T2 hyperintensity (T2L).

IV. To evaluate if participants who receive treatment with standard radiation and temozolomide exhibit a reduction in hyperpolarized 13C lactate/pyruvate or 13C glutamate/pyruvate at post-radiation follow-up compared to their baseline scan. A second group of twenty participants will be studied at the time determined from the prior group to provide the maximum contrast between lactate/pyruvate or glutamate/pyruvate in the lesion versus normal brain.

OUTLINE: Participants are assigned to 1 of 2 cohorts.

COHORT I: Participants receive one or two hyperpolarized carbon C 13 pyruvate injections intravenously (IV) and undergo MRI.

COHORT II: Participants receive hyperpolarized carbon C 13 pyruvate IV and undergo MRI before treatment and 4 weeks after completion of treatment.

After completion of study treatment, participants are followed for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

For Participants in Cohort 1: Histologically proven glioma who have evidence of evaluable disease based on a prior magnetic resonance (MR) scan.

For Participants in Cohort 2: Histologically proven glioma who will be undergoing treatment.

To be included in the study all subjects must also meet the following criteria:

1. Participants must be > 18 years old and with a life expectancy > 12 weeks.
2. Participants must have a Karnofsky performance status of ≥ 60.
3. Participants must have adequate renal function (creatinine < 1.5 mg/dL) before starting therapy. This tests must be performed within 60 days prior to Hyperpolarized Imaging scan.
4. Participants must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy, would compromise the patient's ability to tolerate the imaging examination or any disease that will obscure toxicity or dangerously alter response to the imaging agent.
5. Participants must not have New York Heart Association (NYHA) Grade II or greater congestive heart failure
6. Participants must not have a history of myocardial infarction or unstable angina within 12 months prior to study enrollment.
7. This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. Minorities will actively be recruited to participate. No exclusion to this study will be based on race.
8. Participants must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must sign an authorization for the release of their protected health information.
9. Participants may not be known to be human immunodeficiency virus (HIV)-positive. HIV testing is not required for study participation.
10. Participants must not have a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off all therapy for that disease for a minimum of 3 years.
11. Participants must not be pregnant or breast feeding. Women of childbearing potential are required to obtain a negative pregnancy test within 14 days of Hyperpolarized Imaging scan. Effective contraception (men and women) must be used in subjects of child-bearing potential.

Exclusion Criteria:

1. Participants must be excluded from participating in this study if they are not able to comply with study and/or follow-up procedures.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2015-12-09 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 24 months
  Adverse events will be monitored from just before investigational medicinal product (IMP) administration until the end of study participation. Vital signs (blood pressure and heart rate only) will be recorded at baseline and 30 minutes post injection. For blood pressures and heart rate recorded after IMP administration, the following safety endpoints will be summarized for each part of the study: (1) The occurrence of changes from baseline, at each post-administration time point, greater than a pre-specified magnitude (20 mm Hg for systolic blood pressure, 10 mm Hg for diastolic blood pressure, 10 beats per minute for heart rate). (2) The occurrence of post-administration values outside the normal limits. Toxicities will be graded using the National Cancer Institute (NCI) Common Terminology (Toxicity) Criteria for Adverse Events (CTCAE) version 4.0
Peak lactate/pyruvate ratio in brain tissue | Up to 24 months
  The lactate/pyruvate ratio and/or glutamate/pyruvate will be compared in tumor versus normal appearing brain tissue. Comparisons will be made using a Wilcoxon signed rank test.
Peak lactate/pyruvate ratio in (13C) pyruvate scan | Up to 4 months.
  The lactate/pyruvate ratio and/or glutamate/pyruvate from baseline will be compared to the ratio on the post-radiation therapy (RT) repeat scan. Comparisons will be made using a Wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Chang, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Autry AW, Gordon JW, Chen HY, LaFontaine M, Bok R, Van Criekinge M, Slater JB, Carvajal L, Villanueva-Meyer JE, Chang SM, Clarke JL, Lupo JM, Xu D, Larson PEZ, Vigneron DB, Li Y. Characterization of serial hyperpolarized 13C metabolic imaging in patients with glioma. Neuroimage Clin. 2020;27:102323. doi: 10.1016/j.nicl.2020.102323. Epub 2020 Jun 24. PMID 32623139

DOCUMENTS (1):
  • Informed Consent Form (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/11/NCT03739411/ICF_000.pdf